CLINICAL TRIAL: NCT03535675
Title: A Randomized Double-Blind, Placebo-Controlled Study Of The Effects Of MPX Capsules On Rising Prostate-Specific Antigen Levels In Alanine/Alanine SOD2 Genotype Men Following Initial Therapy For Prostate Cancer
Brief Title: Muscadine Plus (MPX) In Men With Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated by DSMB due to futility.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Greater Washington Community Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: J1823; IRB00166021 (Other: JHM IRB)
Record Dates: First submitted 2018-05-10; First posted 2018-05-24 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Adenocarcinoma of the Prostate

STUDY DESIGN:
Intervention Model Description: This is a multicenter, double-blind, randomized study to evaluate the benefit of MPX supplementation in the subset of men who display the Alanine/Alanine SOD2 genotype of MnSOD. Based on a previous randomized phase II trial of MPX at Hopkins, PSA doubling time (PSA-DT) was prolonged in this subgroup of men.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Muscadine Plus (Experimental): Each treatment cycle consists of once daily oral dosing of 4000 mg Muscadine Plus, every day throughout each 12 week (84 day) cycle. Patients may continue to receive additional cycles of study drug and will be followed every three months with standard visits with their physician until completion of 48 weeks of study treatment, disease progression, or until they wish to discontinue the drug.
  Interventions: Drug: Muscadine Plus
- Placebo (Experimental): Each treatment cycle consists of once daily oral dosing of 4000 mg placebos, every day throughout each 12 week (84 day) cycle. Patients may continue to receive additional cycles of placebo and will be followed every three months with standard visits with their physician until completion of 48 weeks of study treatment, disease progression, or until they wish to discontinue the drug.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Muscadine Plus — Ellagic acid inhibits DNA Methyltransferase. DNA Methyltransferases (DNMTs) are a family of enzymes that regulate chromatin methylation and use S-adenosyl methionine (SAM) as the methyl donor. Ellagic acid's metabolite, urolithin-A inhibits the protein complex nuclear factor kappa-light-enhancer of activated B-cells (NFkB), potentially leading to increased rates of apoptosis and decreases in cancer cell proliferation. Extracts from Vitis rotundifolia have shown inhibition of the phosphatidylinositol 3-kinase-Akt pathway.
  Other Names: MPX
  Arms: Muscadine Plus
Drug: Placebos — The placebo capsules are rice flour that will be placed in white opaque capsules identical to the ones used for MPX.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This research is being done to determine if men with rising PSA after initial therapy for localized prostate cancer who display the Alanine/Alanine SOD2 genotype of MnSOD and supplement their diet with MPX have greater decrease in PSA slope following treatment compared to men that do not supplement with MPX.

DETAILED DESCRIPTION:
Prostate specific antigen (PSA) is a single-chain glycoprotein produced by the epithelial cells of the prostate. PSA has been used for early detection and monitoring of patients with prostate cancer who receive a variety of treatments. Due to the widespread use of serum PSA to monitor for prostate cancer recurrence following primary treatment, there exists a group of men with a rising PSA as their only evidence of recurrence. These patients may not demonstrate clinical or radiographic evidence of disease progression for an average 8 years from the time of detectable PSA to detectable metastatic disease by standard imaging. Currently there are limited treatment options for these patients that may delay disease progression or improve survival, including salvage radiation for prior surgical patients, hormonal therapy, and active surveillance.

Although some surgical patients are candidates for salvage radiation, not all patients will want salvage radiation. Even the early initiation of hormonal therapy (e.g., luteinizing hormone releasing hormone (LHRH) analogs) has not demonstrated a survival benefit, although Schroder et al suggests an advantage for early hormone therapy in the setting of metastatic regional lymph nodes. Furthermore, early initiation of androgen ablation is associated with significant morbidity and impact on quality of life, including fatigue, hot flashes, loss of libido, decreased muscle mass, and osteoporosis with long term use. This group of relatively well men with biochemical recurrence are currently offered androgen ablation therapy or active surveillance (regular PSA monitoring and annual scans) until there is evidence of metastatic disease, because other options have not been available. These patients are excellent candidates for innovative treatments hypothesized to slow the progression of clinical prostate cancer and delay the development of metastatic disease.

As the previous section documents, preclinical studies of muscadine grape skin offer evidence that it may extend the time between biochemical recurrence and development of metastatic disease. While the Phase II study described above found no significant difference in PSA doubling time between placebo and either dose of MPX, there was a signal of benefit in the subgroup analysis of men with the Alanine/Alanine superoxide dismutase 2 (SOD2) genotype that received high dose MPX. It is therefore proposed to test the benefits of high dose MPX in capsule formulation in a randomized, controlled study of men who have failed primary therapy, either radiation, surgery or cryotherapy, as primary treatment for prostate cancer. Eligible subjects will have a rising PSA and will have 3 PSA values at least 7 days apart with a recovered testosterone to be able to calculate a baseline PSA doubling time. The primary endpoint of this study will be mean PSA slope during the study period.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following conditions are eligible for registration and participation in the study:

1. Subject has histologically or cytologically confirmed adenocarcinoma of the prostate
2. Subject has undergone definitive treatment (surgery, surgery with radiation therapy, cryotherapy, radiation therapy or brachytherapy) for the primary prostate tumor (prior chemotherapy is not allowed) .

   a. A subject with a rising PSA post-prostatectomy should consider radiation as a potentially curative alternative. If subject declines radiation or is not a candidate for radiation, he may be considered eligible in this setting.
3. Subject has a rising PSA on a minimum of 3 time points (2 rises) within the 12 months prior to study initiation (this will include the PSA measurement taken at the screening visit, but not at the baseline day 0 study visit).

   For purposes of calculating PSA doubling time (PSADT):
   1. All PSA values used in the calculation should be ≥ 0.20 ng/ml and overall should follow a rising trend;
   2. Record every available PSA drawn within the last 12 months of the most recent local PSA;
   3. The minimum requirement is 3 PSA values obtained over 3 months with a minimum of 4 weeks between measurements;
   4. If there are 4 or more PSAs available, the time interval between the first and last PSA measurements must be at least 3 months, and, there is no minimum time interval requirement between any two PSA measurements;
   5. For radiotherapy only patients, record PSA nadir value and collection date. PSADT (PSA doubling time) must be positive according to Memorial Sloan Kettering Cancer Center Prostate Cancer Nomograms under this link: http://www.mskcc.org/applications/nomograms/prostate/PsaDoublingTime.aspx
4. One of the following criteria must be met.

   1. Absolute level of PSA >0.4 ng/mL following surgery. (surgery only)
   2. Absolute level of PSA >0.4 ng/mL for subjects treated with multiple treatment modalities (e.g., surgery + radiation, surgery + cryotherapy, etc.).
   3. A rise by 2 ng/mL or more above the nadir PSA will be considered the standard definition for biochemical failure after radiation therapy with or without hormonal therapy. (radiation only)
5. Subject is >18 years of age.
6. Subject has life expectancy of greater than 12 months.
7. Subject has Eastern Cooperative Oncology Group performance status 0, 1 or 2
8. Subject has testosterone level of ≥1.5 ng/mL at screening.
9. Subject has normal organ and marrow function as defined below:

   1. Leukocytes >3,000/microliter
   2. absolute neutrophil count >1,500/microliter
   3. platelets >100,000/microliter
   4. total bilirubin <1.5 x upper limit of normal except for Gilberts <2.5 x upper limit of normal
   5. aspartate aminotransferase/Alanine transaminase ≤ 2.5 X upper limit of normal
   6. creatinine ≤ 2.5 upper limit of normal
10. Subject agrees to abstain from other commercially available MuscadinePlus (MP) products (Vinetra, MuscadinePlus or MP capsules) while participating in this study.
11. Subject's use of other dietary/herbal supplements (e.g. saw palmetto, selenium, pomegranate juice or pills, acai concentrated extract, etc) has been stable for at least 2 months prior to screening and the subject agrees not to stop or change the dose(s) while participating in the study.
12. Subject has signed a written informed consent document and agrees to comply with requirements of the study.
13. CT or MRI chest/abdomen/pelvis and bone scan without evidence of metastatic disease as an inclusion.
14. Subject agrees to genotyping of manganese-dependent superoxide dismutase 2 (MnSOD2) gene and any genetic counseling. Only those with Alanine/Alanine SOD2 genotype will be randomized.

Exclusion Criteria:

Subjects meeting the following conditions are not eligible for participation in the study:

1. Subject has known radiographic evidence of metastatic disease, except for presence of positive lymph nodes from the surgical pathology. Pelvic/intraperitoneal lymph nodes less than 1.5 cm maybe considered nonspecific and the patient would be eligible. If there is any clinical suspicion for metastatic disease, CT and Bone Scan must be performed to rule out metastatic disease, within the last four months, per standard of care.
2. Subject has received any therapies that modulate testosterone levels (e.g., androgen ablative/anti-androgen therapy, 5 alpha reductase inhibitors) for a minimum of 12 months prior to study.
3. Subject has had prior or concomitant treatment with experimental drugs, high dose steroids, or any other cancer treatment within 4 weeks prior to the first dose of the study product.
4. Subject has consumed any Muscadine Plus over the past 2 months.
5. Subject has a known allergy to muscadine grapes, ellagic acid or rice
6. Subject has uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Subject has negative PSA doubling time (negative doubling time corresponds with decreasing PSA) Doubling time may be computed using the Sloan Kettering prediction tools posted at http://www.mskcc.org/applications/nomograms/prostate/PsaDoublingTime.aspx

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Channing Paller, M.D, Principal Investigator — SKCCC at Johns Hopkins
Locations (13):
- United States (13):
  - City of Hope, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mandl A, Zahurak ML, Metri NA, Shore ND, Mao S, McKay RR, Taplin ME, Szmulewitz RZ, Maughan BL, Reichert ZR, Kessler ER, Heath EI, Dreicer R, Stein CA, Milne GL, Sfanos KS, Ernst SE, Mummert LA, Cruz-Lebron A, Michel SLJ, Kane MA, Hursey M, Worth MA, Wagner WD, Eshleman JR, Debeljak M, Xu L, Cao H, Dowling D, Marshall CH, Markowski MC, Denmeade SR, Eisenberger MA, Antonarakis ES, Carducci MA, Paller CJ. Muscadine Grape Skin Extract in Biochemically Recurrent Prostate Cancer: A Randomized, Placebo-Controlled, Biomarker-Enriched Trial in Patients With the SOD2 Ala/Ala Variant. Prostate. 2025 Jul;85(10):966-976. doi: 10.1002/pros.24903. Epub 2025 May 5. PMID 40325900

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Muscadine Plus | Placebo
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Muscadine Plus | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Median (Full Range); unit: years] | 75 [60 to 92] | 73 [53 to 83] | 74 [53 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 30 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 26 | 28 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 30 | 59
Pre-study PSA slope [Median (Inter-Quartile Range); unit: ng/mL/Month] — Pre-study PSA slope was calculated using all available PSA measurements in the 12 months prior to enrollment, including screening PSA measurement. An analysis of covariance (ANCOVA) was used to assess the difference in MPX and placebo treatment effects, with on-study PSA slope as the independent variable and treatment arm and pre-study PSA slope covariates. The unit of measure for PSA slope is ng/mL/Month.
  ng/mL/Month | 0.11 [0.03 to 0.29] | 0.1 [0.03 to 0.44] | 0.1 [0.03 to 0.44]

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response
Description: To determine if men who display the Alanine/Alanine superoxide dismutase 2 (SOD2) genotype of MnSOD and supplement their diet with MPX have greater changes in PSA slope following treatment compared to men that do not supplement with MPX.
  PSA response will be measured as the change of serum PSA in ng/mL/month, on-study PSA slope for each patient with comparisons between treatment arms adjusted for pre-study PSA slope; on-study PSA slope was calculated from PSA values taken at baseline,12, 24, 36, and 48 weeks, and calculated as the slope of the simple linear regression of the natural log of PSA versus time in ng/mL/month.
Time Frame: baseline,12, 24, 36, and 48 weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL/Month
Arm/Group | Muscadine Plus | Placebo
Number analyzed (Participants) | 29 | 30
ng/mL/Month | 0.106 [0.08 to 0.13] | 0.089 [0.06 to 0.11]

2. Secondary Outcome: PSA Doubling Time
Description: PSA doubling time (PSADT) will be calculated in months by measuring the PSA values within 12 months from start of intervention.
Time Frame: Up to 26 months
Measure: Median (Full Range); unit: months
Arm/Group | Muscadine Plus | Placebo
Number analyzed (Participants) | 29 | 30
months | 6.56 [2.39 to 20.82] | 6.87 [1.57 to 25.48]

3. Secondary Outcome: PSA Objective Response Rate
Description: The number of patients with a decrease in PSA of ≥50%
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Muscadine Plus | Placebo
Number analyzed (Participants) | 29 | 30
Participants | 0 | 0

4. Secondary Outcome: PSA Progression
Description: The time to disease progression for both treatment groups by PSA progression. PSA progression is defined as an increase in PSA greater than 50% and >5 ng/ml above nadir.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Muscadine Plus | Placebo
Number analyzed (Participants) | 29 | 30
months | NA [NA to NA] — The median had not been reached in the MPX arm at the time of the analysis. | 13.77 [11.24 to NA] — The upper limit of confidence interval was not reached.at the time of analysis.

5. Secondary Outcome: Radiographic Progression
Description: The time to disease progression for both treatment groups by radiologic disease progression (i.e. development of metastatic disease).
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Muscadine Plus | Placebo
Number analyzed (Participants) | 29 | 30
months | NA [NA to NA] — There were only two events, so Radiographic progression-free survival (rPFS) could not be calculated. | NA [NA to NA] — There were only two events, so Radiographic progression-free survival (rPFS) could not be calculated.

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Muscadine Plus | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/29 | 6/30
Other Adverse Events (participants affected / at risk) | 22/29 | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Muscadine Plus (N=29) | Placebo (N=30)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Muscadine Plus (N=29) | Placebo (N=30)
flatulence (Gastrointestinal disorders) | 1 (3) | 1 (3)
constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 2 (4) | 2 (4)
pain (General disorders) | 1 (2) | 0 (0)
edema limbs (General disorders) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
localized edema (General disorders) | 0 (0) | 1 (1)
dysuria (Renal and urinary disorders) | 1 (1) | 1 (3)
hematuria (Renal and urinary disorders) | 1 (2) | 1 (2)
urinary frequency (Renal and urinary disorders) | 1 (2) | 0 (0)
urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
shingles (Infections and infestations) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (2)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 1 (1) | 1 (2)
peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
spasticity (Nervous system disorders) | 1 (1) | 0 (0)
creatinine increased (Investigations) | 1 (2) | 1 (1)
white blood cell decreased (Investigations) | 0 (0) | 2 (2)
aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
hot flashes (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03535675/Prot_SAP_001.pdf